CLINICAL TRIAL: NCT05385185
Title: Clinical Observation of ICI Combined With Recombinant Human Endostatin on Leptomeningeal Metastasis of Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Hui Bu, The department of neurology, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH006
Record Dates: First submitted 2021-07-07; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Leptomeningeal Metastasis; Immune Checkpoint Inhibitor; Endostatin
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — camrelizumab; envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leptomeningeal metastases received PD-1 inhibitor and recombinant human endostatin (Experimental): Camrelizumab 200mg intravenously, once every 21 days or envafolimab 150mg subcutaneous injection,once a week Endostatin 30mg/d was administered intravenously for 7 days (d1-d7). The interval between Endostatin and next was 2 weeks.
  Interventions: Drug: Camrelizumab or envafolimab

INTERVENTIONS:
Drug: Camrelizumab or envafolimab — combine Camrelizumab or envafolimab with Recombinant human vascular endostatin
  Other Names: Recombinant human vascular endostatin

SUMMARY:
immune checkpoint inhibitor combined with recombinant human endostatin can improve the 3-month OS rate of leptomeningeal metastasis of lung cancer, and the combination is safe

DETAILED DESCRIPTION:
We will recruit 20 patients with leptomeningeal metastases from lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender unlimited;
2. A clear diagnosis of leptomeningeal metastases derived from lung cancer , including positive cerebrospinal fluid cytology and/or neuroimaging diagnosis;
3. A clear history of lung cancer, including histopathological diagnosis, or a combination of cytopathology and imaging;
4. Proper organ function (neutrophil count ≥1.5× 109 /L, platelet count ≥100× 109 /L, hemoglobin concentration ≥90g/L, serum transaminase concentration ≤2.5 times the limit of normal value, serum creatinine concentration ≤ 1.5 times the upper limit of normal value, proteinuria ≤1+)
5. Dexamethasone ≤2 mg (or equivalent) 7 days before the start of treatment in patients requiring long-term use of the hormone
6. Signed the informed consent and was willing to follow the experimental protocol and follow-up

Exclusion Criteria:

1. Patients with positive driver genes and effective treatment, such as patients with positive EGFR gene sensitive mutation
2. Severe infections or serious comorbidities, such as hemorrhagic peptic ulcer, intestinal obstruction, heart failure, kidney failure, or poorly controlled diabetes;
3. Be allergic to PD-1 inhibitor and recombinant human endostatin
4. The female patient planned to be pregnant, was pregnant and lactating -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
3-month overall survival rate | 3 month
  The 3-month survival rate after treatment
safty | 2 years
  Adverse events related to treatment

SECONDARY OUTCOMES:
iPFS | 2 years
  Intracranial progression-free survival
extracranial PFS | 2 years
  extracranial progression-free survival
DCR | 2 years
  disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Hebei, China

IPD SHARING:
Plan to Share IPD: No
the patients information should be protected